CLINICAL TRIAL: NCT05580302
Title: Cortical Silent Period in Laryngeal Dystonia
Acronym: cSPDystonia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Split, School of Medicine (Other)
Collaborators: University Hospital of Split (Other)
Responsible Party: Principal Investigator, Maja Rogić Vidaković, Research Associate, University of Split, School of Medicine
Other Study IDs: 003-08/22-03/0003
Record Dates: First submitted 2022-10-10; First posted 2022-10-14 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Laryngeal Dystonia; Spasmodic Dysphonia
Keywords: laryngeal dystonia; cortical silent period; spasmodic dysphonia; transcranial magnetic stimulation
MeSH Terms: conditions — Dysphonia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Laryngeal Dystonia: The study will be performed on 10-15 (maximal 20) subjects with diagnosed laryngeal dystonia who meet the exclusion/ inclusion criteria.
  Inclusion criteria: adults (18-65 years old) who have confirmed diagnosis of laryngeal dystonia, no implanted metals in body (e.g. pacemaker, metal prosthesis in skull and oral cavity).
  Exclusion criteria: pregnancy, other neurological disorders, psychiatric disorders, epilepsy or history of previous epilepsy attack, using of brain affecting pharmaceuticals, traumatic, tumor, infectious, metabolic brain lesions, heart conditions (15 ).
  The composition of the group is represented is both gender, various age gap, and different height.
  Before the beginning of testing, all subjects with a confirmed diagnosis of laryngeal dystonia will be once again evaluated by a specialist otorhinolaryngologist at the University Hospital of Split. Medical documentation of the examination will be available for further analysis.
  Interventions: Other: Transcranial Magnetic Stimulation (TMS)
- Healthy subjects: The study will be performed on 20 healthy volunteering subjects who meet the exclusion/ inclusion criteria.
  Inclusion criteria: healthy adults (18-65 years old), no implanted metals in body (e.g. pacemaker, metal prosthesis in the skull and oral cavity) Exclusion criteria: pregnancy, neurological disorders, psychiatric disorders, epilepsy or history of previous epilepsy attack, using of the brain affecting pharmaceuticals, traumatic, tumor, infectious, metabolic brain lesions, heart conditions.
  The composition of the group is represented is both gender, various age gap, and different height.
  Interventions: Other: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Other: Transcranial Magnetic Stimulation (TMS) — An anatomical T1 magnetic resonance image (MRI) with high resolution will be acquired on a separate day before the TMS experiment. The image will be imported into the neuronavigation system (Nexstim, Helsinki, Finland) to guide the localization of the primary motor cortex (M1) for laryngeal muscle representation. Prior to M1 mapping for laryngeal muscle representation, mapping of the representation for hand muscle representation will be performed. Hand region excitability (abductor pollicis brevis, APB) will be evaluated by using surface electrodes attached to the right-hand APB muscle. The cSP threshold is defined as the lowest TMS intensity that elicits a cSP in 5 out of 10 consecutive trials. Single-pulse cortical stimulations will be performed during the vocalization of sustained /i/ sound.

SUMMARY:
The goal of this observational study is to evaluate the cortical silent period (cSP) in cricothyroid muscle (CT) in laryngeal dystonia and control healthy subjects. The study will provide norms related to latency and amplitude of motor evoked potentials (MEPs) and duration of cSP in CT muscle in laryngeal dystonia and control healthy subjects.

Findings may give a baseline in comparison to findings in laryngeal diseases and insight into maladaptive cortical control function during phonation in laryngeal diseases like laryngeal dystonia.

DETAILED DESCRIPTION:
Transcranial magnetic stimulation (TMS)-induced cSP provide a noninvasive "in vivo" insight into how the human motor cortical inhibitory pathway function by generating electric current at a specific brain area through electromagnetic induction. The stimulator generates a changing electric current within the coil, which induces a magnetic field that then causes a second inductance of inverted electric charge within the brain itself. A single supra-threshold pulse of TMS over the human motor cortex elicits multiple descending volleys (I-waves) that generate a motor evoked potential (MEP) followed by a period of electromyographic silence in the tonically contracted target muscle (cSP). To date, methodologies for mapping the primary motor cortex (M1) with TMS and intraoperatively by electrical stimulation techniques have been previously developed to record corticobulbar motor evoked potentials (MEP) from laryngeal muscles. Except for estimating the amplitude and latency of MEPs recorded from laryngeal muscles, the cSP was investigated from thyroarytenoid muscle (TA) as a measure of M1 excitability in the TMS study. Previous work using TMS has indicated reduced inhibition to be characteristic of focal laryngeal dystonia. According to investigators' knowledge, cSP from other laryngeal muscles other than TA has not been investigated so far.

The proposed study analyses neurophysiological CNS data, including motor evaluation of corticospinal and corticobulbar pathways by recording MEPs and cSP using TMS.

Firstly, a questionnaire will be given to check for any previous neurological conditions, and subjects will provide signatures on participation in the study. The MRI of the subject's brain will be performed, and then 3D reconstructed for the use of TMS. The evaluation of the MRI will be done by radiologists at University Hospital Split. With the subject comfortably seated, the MRI is co-registered to the subject's head using the tracking system with TMS's unique forehead tracker. After TMS measurement of the MEP and cSP of CT muscle of individual subjects will be recorded. Data collected will be analyzed using MATLAB 2022a (MathWorks, USA). Measurements and data evaluation will be performed at the School of Medicine University in Split.

An otorhinolaryngology specialist will be consulted for the correct placement of the recording electrodes (Hookwire IOM electrodes, disposable subdermal needle electrode, 0.4 x 13 mm, SGM d.o.o, G. Novaka 22 a, 21000 Split, Croatia) into the CT muscle.

ELIGIBILITY:
Inclusion Criteria:

* adults (18-65 years old), no implanted metals in the body (e.g. pacemaker, metal prosthesis in the skull and oral cavity).

Exclusion Criteria:

* pregnancy, other neurological disorders (except laryngeal dystonia in the laryngeal dystonia group), psychiatric disorders, epilepsy or history of previous epilepsy attack, using of brain-affecting pharmaceuticals, traumatic, tumor, infectious, metabolic brain lesions, heart conditions.

The composition of the group is represented is both gender, various age gap, and different height.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Inclusion Criteria:
  * adults (18-65 years old) with diagnosed laryngeal dystonia, no implanted metals in the body (e.g. pacemaker, metal prosthesis in the skull and oral cavity).
  Exclusion Criteria:
  * pregnancy, other neurological disorders, psychiatric disorders, epilepsy or history of previous epilepsy attack, use of brain-affecting pharmaceuticals, traumatic, tumor, infectious, metabolic brain lesions, heart conditions.
  The composition of the group is represented is both gender, various age gap, and different height.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Motor evoked potential (MEP) latency | MEP latency evaluated on the first day of the arrival on TMS experiment
  MEP latency is expressed in milliseconds
Motor evoked potential (MEP) amplitude | MEP amplitude evaluated on the first day of the arrival on TMS experiment
  MEP amplitude is expressed in microvolts
Duration of cortical silent period (cSP) | cSP duration evaluated on the first day of the arrival on TMS experiment
  cSP is expressed in milliseconds

CONTACTS AND LOCATIONS:
Overall Officials: Maja Rogić Vidaković, PhD, Principal Investigator — University of Split, School of Medicine
Locations (1):
- University of Split School of Medicine, Split, Croatia

IPD SHARING:
Plan to Share IPD: Undecided
Upon request.

REFERENCES:
- [Background] Blitzer A, Brin MF, Stewart CF. Botulinum toxin management of spasmodic dysphonia (laryngeal dystonia): a 12-year experience in more than 900 patients. Laryngoscope. 2015 Aug;125(8):1751-7. doi: 10.1002/lary.25273. No abstract available. PMID 26200329
- [Background] Pirio Richardson S, Wegele AR, Skipper B, Deligtisch A, Jinnah HA; Dystonia Coalition Investigators. Dystonia treatment: Patterns of medication use in an international cohort. Neurology. 2017 Feb 7;88(6):543-550. doi: 10.1212/WNL.0000000000003596. Epub 2017 Jan 11. PMID 28077492
- [Background] Deletis V, Rogic M, Fernandez-Conejero I, Gabarros A, Jeroncic A. Neurophysiologic markers in laryngeal muscles indicate functional anatomy of laryngeal primary motor cortex and premotor cortex in the caudal opercular part of inferior frontal gyrus. Clin Neurophysiol. 2014 Sep;125(9):1912-22. doi: 10.1016/j.clinph.2014.01.023. Epub 2014 Feb 11. PMID 24613682
- [Background] Chen M, Summers RL, Goding GS, Samargia S, Ludlow CL, Prudente CN, Kimberley TJ. Evaluation of the Cortical Silent Period of the Laryngeal Motor Cortex in Healthy Individuals. Front Neurosci. 2017 Mar 7;11:88. doi: 10.3389/fnins.2017.00088. eCollection 2017. PMID 28326007
- [Background] Chen M, Summers RLS, Prudente CN, Goding GS, Samargia-Grivette S, Ludlow CL, Kimberley TJ. Transcranial magnetic stimulation and functional magnet resonance imaging evaluation of adductor spasmodic dysphonia during phonation. Brain Stimul. 2020 May-Jun;13(3):908-915. doi: 10.1016/j.brs.2020.03.003. Epub 2020 Mar 13. PMID 32289724
- [Background] Rossini PM, Burke D, Chen R, Cohen LG, Daskalakis Z, Di Iorio R, Di Lazzaro V, Ferreri F, Fitzgerald PB, George MS, Hallett M, Lefaucheur JP, Langguth B, Matsumoto H, Miniussi C, Nitsche MA, Pascual-Leone A, Paulus W, Rossi S, Rothwell JC, Siebner HR, Ugawa Y, Walsh V, Ziemann U. Non-invasive electrical and magnetic stimulation of the brain, spinal cord, roots and peripheral nerves: Basic principles and procedures for routine clinical and research application. An updated report from an I.F.C.N. Committee. Clin Neurophysiol. 2015 Jun;126(6):1071-1107. doi: 10.1016/j.clinph.2015.02.001. Epub 2015 Feb 10. PMID 25797650
- [Background] Simonyan K, Barkmeier-Kraemer J, Blitzer A, Hallett M, Houde JF, Jacobson Kimberley T, Ozelius LJ, Pitman MJ, Richardson RM, Sharma N, Tanner K; The NIH/NIDCD Workshop on Research Priorities in Spasmodic Dysphonia/Laryngeal Dystonia. Laryngeal Dystonia: Multidisciplinary Update on Terminology, Pathophysiology, and Research Priorities. Neurology. 2021 May 25;96(21):989-1001. doi: 10.1212/WNL.0000000000011922. Epub 2021 Apr 15. PMID 33858994
- [Background] Rogic Vidakovic M, Schonwald MZ, Rotim K, Juric T, Vulevic Z, Tafra R, Banozic A, Hamata Z, Dogas Z. Excitability of contralateral and ipsilateral projections of corticobulbar pathways recorded as corticobulbar motor evoked potentials of the cricothyroid muscles. Clin Neurophysiol. 2015 Aug;126(8):1570-7. doi: 10.1016/j.clinph.2014.11.001. Epub 2014 Nov 8. PMID 25481338